CLINICAL TRIAL: NCT00469131
Title: Randomized Comparative Study on Effects of Immunosuppression on HCV Recurrence After Living Donor Liver Transplantation - Comparison Between Tacrolimus + MMF and Tacrolimus + Steroid
Brief Title: Effects of Immunosuppression on HCV Recurrence After Living Donor Liver Transplantation - Comparative Study Between Tacrolimus + MMF and Tacrolimus + Steroid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Kyoto University (Other)
Responsible Party: Shinji Uemoto, M.D. PhD, Professor of Department of Hepatobiliary Pancreatic Surgery and Transplantation, Kyoto University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHA-LD-03-01
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Hepatitis C; Liver Cirrhosis
Keywords: liver transplantation,; HCV recurrence,; immunosuppression
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis | interventions — Tacrolimus; Steroids; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Drug: (Active Comparator): tacrolimus + steroid
  Interventions: Drug: tacrolimus + steroid
- 2 Drug: (Active Comparator): tacrolimus + mycophenolate mofetil
  Interventions: Drug: tacrolimus + mycophenolate mofetil

INTERVENTIONS:
Drug: tacrolimus + steroid
  Arms: 1 Drug:
Drug: tacrolimus + mycophenolate mofetil
  Arms: 2 Drug:

SUMMARY:
The aim of this study is to compare immunosuppression protocol of tacrolimus + MMF with that of tacrolimus + steroid for preventing recurrence of hepatitis C after living donor liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of living donor liver transplantation for HCV-related cirrhosis

Exclusion Criteria:

* ABO blood type incompatible transplant case
* Renal dysfunction (serum creatinine >2.0 mg/dL)
* WBC < 1,000/mm3
* Hemoglobin < 8 g/dL
* Platelet <30,000 /mm3

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2003-09; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Event-free survival time at the end of first year after living liver transplantation. | 1 year

SECONDARY OUTCOMES:
HCV-RNA value, patient survival, recurrence-free survival, rate of interferon therapy induction, rate of steroid pulse for rejection, chronic rejection | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shinji Uemoto, MD, PhD, Principal Investigator — Kyoto University Hospital
Locations (1):
- Kyoto University Hospital, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Takada Y, Kaido T, Asonuma K, Sakurai H, Kubo S, Kiuchi T, Inomata Y, Isaji S, Tsumura H, Teramukai S, Matsubara Y, Sakabayashi S, Uemoto S. Randomized, multicenter trial comparing tacrolimus plus mycophenolate mofetil to tacrolimus plus steroids in hepatitis C virus-positive recipients of living donor liver transplantation. Liver Transpl. 2013 Aug;19(8):896-906. doi: 10.1002/lt.23679. PMID 23696054